CLINICAL TRIAL: NCT02302807
Title: A Phase III, Open-Label, Multicenter, Randomized Study to Investigate the Efficacy and Safety of Atezolizumab (Anti-PD-L1 Antibody) Compared With Chemotherapy in Patients With Locally Advanced or Metastatic Urothelial Bladder Cancer After Failure With Platinum-Containing Chemotherapy
Brief Title: A Study of Atezolizumab Compared With Chemotherapy in Participants With Locally Advanced or Metastatic Urothelial Bladder Cancer [IMvigor211]
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29294; 2014-003231-19 (EudraCT Number)
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Results first posted 2018-04-11 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — atezolizumab; Docetaxel; Paclitaxel; vinflunine

ARMS (2):
- Arm A: Atezolizumab (Experimental): Atezolizumab will be administered intravenously at a fixed dose of 1200 milligrams (mg) on Day 1 of each 21-day cycle. Participants will receive atezolizumab as long as they continue to experience clinical benefit in the opinion of the investigator until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator.
  Interventions: Drug: Atezolizumab (MPDL3280A) [TECENTRIQ], an engineered anti-PDL1 antibody
- Arm B: Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) (Active Comparator): Participants randomized to the chemotherapy arm will receive vinflunine, paclitaxel, or docetaxel per the investigator's choice. Vinflunine 320 milligrams per square meter (mg/m^2), paclitaxel 175 mg/m^2, or docetaxel 75 mg/m^2 will be administered intravenously on Day 1 of each 21-day cycle until disease progression per standard RECIST v1.1 or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Paclitaxel; Drug: Vinflunine

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A) [TECENTRIQ], an engineered anti-PDL1 antibody — Atezolizumab will be administered intravenously at a fixed dose of 1200 mg on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
  Arms: Arm A: Atezolizumab
Drug: Docetaxel — Docetaxel 75 mg/m^2 will be administered intravenously on Day 1 of each 21-day cycle.
  Arms: Arm B: Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel)
Drug: Paclitaxel — Paclitaxel 175 mg/m^2 will be administered intravenously on Day 1 of each 21-day cycle.
  Arms: Arm B: Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel)
Drug: Vinflunine — Vinflunine 320 mg/m^2 will be administered intravenously on Day 1 of each 21-day cycle.
  Arms: Arm B: Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel)

SUMMARY:
This is a Phase III, global, multicenter, open-label, two-arm, randomized, controlled study designed to evaluate the efficacy and safety of atezolizumab compared with chemotherapy in participants with locally advanced or metastatic urothelial bladder cancer (UBC) who have progressed during or following a platinum-containing regimen. The anticipated time on study treatment is based on continued clinical benefit, i.e., until disease progression or unacceptable toxicity. The target sample size is 931 participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic UBC (including renal pelvis, ureters, urinary bladder, and urethra).
* Representative tumor specimens as specified by the protocol
* Disease progression during or following treatment with at least one platinum-containing regimen for inoperable, locally advanced or metastatic UBC or disease recurrence
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than or equal to (>/=) 12 weeks
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end organ function
* For women of childbearing potential, agreement to refrain from heterosexual intercourse or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 5 months after the last dose of atezolizumab, 3 months after the last dose of vinflunine and 6 months from the last dose of paclitaxel or docetaxel.
* For men, agreement to refrain from heterosexual intercourse or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 3 months after the last dose of vinflunine and 6 months from the last dose of paclitaxel or docetaxel, and agreement to refrain from donating sperm

Exclusion Criteria:

* Any approved anti-cancer therapy within 3 weeks prior to initiation of study treatment
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment
* Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments
* Leptomeningeal disease
* Malignancies other than UBC within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome, or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer
* Pregnant and lactating women
* Significant cardiovascular disease
* Severe infections within 4 weeks prior to randomization
* Major surgical procedure other than for diagnosis within 4 weeks prior to randomization
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins; known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease
* Prior allogeneic stem cell or solid organ transplant
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Positive test for human immunodeficiency virus (HIV) and/or active hepatitis B or hepatitis C or tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks prior to randomization
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies, including anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1) or anti-programmed death-ligand 1 (anti-PD-L1) therapeutic antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 931 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (217):
- United States (6):
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Emory University; Winship Cancer Institute, Atlanta, Georgia
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Duke Cancer Center, Durham, North Carolina
  - Bon Secours - St. Francis Hospital, Greenville, South Carolina
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
- Australia (4):
  - Royal Brisbane and Women's Hospital; Medical Oncology, Herston, Queensland
  - Royal Adelaide Hospital; Oncology, Adelaide, South Australia
  - Monash Medical Centre; Oncology, Clayton, Victoria
  - Austin and Repatriation Medical Centre; Cancer Services, Melbourne, Victoria
- Austria (2):
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Abt. für Onkologie, Vienna
  - Kaiser-Franz-Josef-Spital; Zent.Onkologie und Hamatologie, Vienna
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Canada (11):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Bcca - Cancer Center Southern Interior, Kelowna, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Bcca - Vancouver Island Cancer Centre; Oncology, Victoria, British Columbia
  - Royal Victoria Hospital, Barrie, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - Sault Area Hospitals, Sault Ste. Marie, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
- Czechia (5):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - MULTISCAN, s.r.o., Radiologicke centrum Pardubice, Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- Denmark (2):
  - Herlev Hospital; Onkologisk afdeling, Herlev
  - Rigshospitalet; Onkologisk Klinik, København Ø
- Finland (2):
  - Docrates Cance Center, Helsinki
  - Turku University Central Hospital; Urology clinic, Turku
- France (25):
  - Ico - Paul Papin, Angers
  - Institut Sainte Catherine;Recherche Clinique, Avignon
  - Chr De Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Francois Baclesse; Recherche Clinique, Caen
  - CHU Henri Mondor; Service d'Oncologie Medicale, Créteil
  - Clinique Chenieux; Oncology, Limoges
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut J Paolii Calmettes, Marseille
  - Institut régional du Cancer Montpellier, Montpellier
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - Centre Antoine Lacassagne, Nice
  - CHU De Nimes, Hopital Caremeau; Service De Neurologie Du Prof. Pierre Labauge, Nîmes
  - Hopital Cochin; Unite Fonctionnelle D Oncologie, Paris
  - Institut Curie; Recherche Clinique, Paris
  - Hopital Saint Louis; Oncologie Medicale, Paris
  - Hopital Europeen Georges Pompidou; Service D'Oncologie Medicale, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - ICO - Site René Gauducheau, Saint-Herblain
  - Hopital Hautepierre; Hematologie Oncologie, Strasbourg
  - Hopital Foch; Oncologie, Suresnes
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif
- Germany (15):
  - Uniklinik RWTH Aachen; Klinik für Urologie, Aachen
  - Charité - Universitätsmedizin Berlin; CC 8: Chirurgische Medizin; Klinik für Urologie, Berlin
  - Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik für Urologie, Dresden
  - Universitätsklinikum Düsseldorf; Urologische Klinik, Düsseldorf
  - Friedrich-Alexander-Universität Erlangen-Nürnberg; Medizinische Klinik V, Erlangen
  - Universitätsklinikum Freiburg; Chirurgische Klinik; Abteilung Urologie, Freiburg im Breisgau
  - Universitätsmedizin Göttingen Georg-August-Universität; Klinik für Urologie, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf Onkologisches Zentrum Medizinische Klinik II, Hamburg
  - Nationales Centrum für Tumorerkrankungen Heidelberg (NCT); Thoraxklinik Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes; Klinik für Urologie und Kinderurologie, Homburg/Saar
  - Universitätsklinikum Magdeburg A.ö.R., Klinik f. Urologie u. Kinderurologie, Magdeburg
  - Medizinische Fakultät Mannheim, Universitätsklinikum Mannheim, Klinik für Urologie, Mannheim
  - Klinikum rechts der Isar der TU München; Urologische Klinik und Poliklinik, München
  - Universitätsklinikum Tübingen; Klinik für Urologie, Tübingen
  - Universitätsklinikum Ulm; Klinik für Urologie, Ulm
- Greece (4):
  - Alexandras General Hospital of Athens; Oncology Department, Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - University Hospital of Patras Medical Oncology, Pátrai
  - Euromedical General Clinic of Thessaloniki; Oncology Department, Thessaloniki
- Hungary (5):
  - Semmelwies University of Medicine; Urology Dept., Budapest
  - Orszagos Onkologiai Intezet; "C" Belgyógyászati-Onkológiai és Klinikai Farmakológiai Osztály, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Kecskemeti Onkoradilogai Centrum, Kecskemét
  - Hetenyi Geza County Hospital; Onkologiai Kozpont, Szolnok
- Italy (13):
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Oncologia, San Giovanni Rotondo, Apulia
  - Azienda Ospedaliera A. Cardarelli; Dip. Oncopneumoematologico, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Oncologia, Modena, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia, Udine, Friuli Venezia Giulia
  - Azienda Ospedaliera San Camillo Forlanini; Oncologia Medica, Rome, Lazio
  - Asst Papa Giovanni XXIII; Oncologia Medica, Bergamo, Lombardy
  - ASST DI CREMONA; Dip. Medicina - S.C. Oncologia, Cremona, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo; Dipartimento Oncologico, Candiolo, Piedmont
  - Casa Di Cura Di Alta Specialita La Maddalena; Dept. Oncologico Di Iii Livello, Palermo, Sicily
  - Azienda USL8 Arezzo-Presidio Ospedaliero 1 San Donato;U.O.C. Oncologia, Arezzo, Tuscany
  - Azienda Ospedaliero-Universitaria Careggi;S.C. Oncologia Medica 1, Florence, Tuscany
- Japan (25):
  - Nagoya University Hospital; Urology, Aichi
  - Hirosaki University School of Medicine & Hospital; Urology, Aomori
  - Chiba Cancer Center; Urology, Chiba
  - National Cancer Center Hospital East; Breast and Medical Oncology, Chiba
  - National Hospital Organization Shikoku Cancer Center; Urology, Ehime
  - Harasanshin Hospital; Urology, Fukuoka
  - Kyushu University Hospital; Urology, Fukuoka
  - Gunma University Hospital; Urology, Gunma
  - Hiroshima City Hiroshima Citizens Hospital; Urology, Hiroshima
  - Sapporo Medical University Hospital; Urology, Hokkaido
  - Hokkaido University Hospital; Urology, Hokkaido
  - University of Tsukuba Hospital; Urology, Ibaraki
  - Yokohama City University Hospital; Urology, Kanagawa
  - Kumamoto University Hospital; Urology, Kumamoto
  - Niigata Cancer Center Hospital;Urology, Niigata
  - Iwate Medical University Hospital; Urology, Numakunai
  - Osaka International Cancer Institute; Urology, Osaka
  - Osaka University Hospital; Urology, Osaka
  - Kindai University Hospital; Urology, Osaka
  - Shizuoka Cancer Center; Urology, Shizuoka
  - Tokushima University Hospital; Urology, Tokushima
  - National Cancer Center Hospital; Urology, Tokyo
  - Toranomon Hospital; Medical Oncology, Tokyo
  - Nippon Medical School Hospital; Urology, Tokyo
  - The Cancer Institute Hospital, JFCR; Urology, Tokyo
- Netherlands (5):
  - The Netherlands Cancer Institute - Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Spaarne Ziekenhuis; Inwendige Geneeskunde, Hoofddorp
  - Maastricht University Medical Centre; Medical Oncology, Maastricht
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Isala Klinieken, Zwolle
- Norway (3):
  - Sørlandet Sykehus Kristiansand, Kristiansand
  - Uni Hospital of Tromso; Dept. of Oncology, Tromsø
  - St. Olavs Hospital; Kreftavdelingen, Trondheim
- Poland (6):
  - Medical University of Bialystok; Oncology clinic, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - COZL Oddzial Onkologii Klinicznej z pododdzialem Chemioterapii Dziennej, Lublin
  - Oddzial Chemioterapii Szpitala Klinicznego Nr 1 w Poznaniu, Poznan
  - Centrum onkologii Instytutu im. Marii Sklodowskiej-Curie; Klinika Nowotworow Ukladu Moczowego, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Miklulicza-Radeckiego we Wrocławiu; Departament Of Urology, Wroclaw
- Portugal (3):
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - Hospital Beatriz Angelo; Departamento de Oncologia, Loures
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Romania (7):
  - Spitalul Judetean de Urgenta Dr Constantin Opris, Baia Mare
  - Institute Of Oncology Bucharest; Medical Oncology, Bucharest
  - Institut Oncologic Ion Chiricuta; Departament Radioterapie, Cluj-Napoca
  - Oncology Center Sf. Nectarie, Craiova
  - Euroclinic Center of Oncology SRL, Iași
  - Spital Clinic Judetean Mures; Oncologie, Târgu Mureş
  - ONCOMED - Medical Centre, Timișoara
- Russia (5):
  - GBUZ Nizhegorodskay Region: Clinical Diagnostic Center, Nizhny Novgorod, Niznij Novgorod
  - Altai Regional Oncological Center, Barnaul
  - Federal State Institution, Moscow Research Oncology Institute n.a. P.A. Hertzen; Oncourology, Moscow
  - St. Petersburg Oncology Hospital, Saint Petersburg
  - SBI of Healthcare of Stavropol region Stavropol Regional Clinical Oncology Dispensary, Stavropol
- Serbia (3):
  - Clinical Center of Serbia; Clinic of Urology, Belgrade
  - Institute for Oncology and Radiology of Serbia; Medical Oncology, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Samsung Medical Center, Seoul
- Spain (19):
  - Hospital Universitario Son Espases; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital de Navarra; Servicio de Oncologia, Navarra, Navarre
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Clinic i Provincial; Servicio de Farmacia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital San Pedro De Alcantara; Servicio de Oncologia, Cáceres
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
  - Hospital Clínico Universitario de Valencia; Servicio de Oncología, Valencia
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset; Jubileumskliniken, Gothenburg
  - Karolinska Hospital; Oncology - Radiumhemmet, Stockholm
  - Norrlands Uni Hospital; Onkologi Avd., Umeå
- Switzerland (5):
  - Inselspital Bern; Universitätsklinik für medizinische Onkologie, Bern
  - Kantonsspital Graubünden;Onkologie und Hämatologie, Chur
  - HUG; Oncologie, Geneva
  - Kantonsspital St. Gallen; Onkologie/Hämatologie, Sankt Gallen
  - UniversitätsSpital Zürich; Zentrum für Hämatologie und Onkologie, Klinik für Onkologie, Zurich
- Taiwan (4):
  - China Medical University Hospital; Urology, Taichung
  - Taichung Veterans General Hospital; Division of Urology, Taichung
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
  - TAIPEI VETERANS GENERAL HOSPITAL, Urology, Taipei
- Turkey (Türkiye) (8):
  - Uludag Uni Hospital; Oncology, Bursa
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Bezmialem Vakif Univ Medical, Istanbul
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
  - Istanbul VKV American Hospital; Medical Oncology, Istanbul
  - Ege Uni Medical Faculty Hospital; Oncology Dept, Izmir
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sıhhiye, Ankara
- United Kingdom (19):
  - University Hospital Birmingham The Cancer Centre, Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Cheltenham General Hospital, Cheltenham
  - University Hospital coventry; Oncology Department, Coventry
  - Royal Devon & Exeter Hospital; Oncology Centre, Exeter
  - Royal Lancaster Infirmary, Morecambe Bay Hospitals Nhs Trust, Lancaster
  - St James Institute of Oncology, Leeds
  - Leicester Royal Infirmary; Dept. of Medical Oncology, Leicester
  - Barts and The London, London
  - Royal Free Hospital; Dept of Oncology, London
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Northern Centre for Cancer Care; Northern Centre for Cancer Care, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Scunthorpe General Hospital; Dept of Oncology, Scunthorpe
  - Southampton General Hospital; Medical Oncology, Southampton
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] van der Heijden MS, Loriot Y, Duran I, Ravaud A, Retz M, Vogelzang NJ, Nelson B, Wang J, Shen X, Powles T. Atezolizumab Versus Chemotherapy in Patients with Platinum-treated Locally Advanced or Metastatic Urothelial Carcinoma: A Long-term Overall Survival and Safety Update from the Phase 3 IMvigor211 Clinical Trial. Eur Urol. 2021 Jul;80(1):7-11. doi: 10.1016/j.eururo.2021.03.024. Epub 2021 Apr 23. PMID 33902955
- [Derived] Shemesh CS, Chan P, Legrand FA, Shames DS, Das Thakur M, Shi J, Bailey L, Vadhavkar S, He X, Zhang W, Bruno R. Pan-cancer population pharmacokinetics and exposure-safety and -efficacy analyses of atezolizumab in patients with high tumor mutational burden. Pharmacol Res Perspect. 2020 Dec;8(6):e00685. doi: 10.1002/prp2.685. PMID 33241650
- [Derived] Morrissey KM, Marchand M, Patel H, Zhang R, Wu B, Phyllis Chan H, Mecke A, Girish S, Jin JY, Winter HR, Bruno R. Alternative dosing regimens for atezolizumab: an example of model-informed drug development in the postmarketing setting. Cancer Chemother Pharmacol. 2019 Dec;84(6):1257-1267. doi: 10.1007/s00280-019-03954-8. Epub 2019 Sep 21. PMID 31542806
- [Derived] Rassy EE, Bakouny Z, Aoun F, Haddad FG, Sleilaty G, Assi T, Kattan J. A network meta-analysis of the PD(L)-1 inhibitors in the salvage treatment of urothelial bladder cancer. Immunotherapy. 2018 Jun;10(8):657-663. doi: 10.2217/imt-2017-0190. Epub 2018 Mar 22. PMID 29562804
- [Derived] Powles T, Duran I, van der Heijden MS, Loriot Y, Vogelzang NJ, De Giorgi U, Oudard S, Retz MM, Castellano D, Bamias A, Flechon A, Gravis G, Hussain S, Takano T, Leng N, Kadel EE 3rd, Banchereau R, Hegde PS, Mariathasan S, Cui N, Shen X, Derleth CL, Green MC, Ravaud A. Atezolizumab versus chemotherapy in patients with platinum-treated locally advanced or metastatic urothelial carcinoma (IMvigor211): a multicentre, open-label, phase 3 randomised controlled trial. Lancet. 2018 Feb 24;391(10122):748-757. doi: 10.1016/S0140-6736(17)33297-X. Epub 2017 Dec 18. PMID 29268948
- [Derived] Balar AV, Galsky MD, Rosenberg JE, Powles T, Petrylak DP, Bellmunt J, Loriot Y, Necchi A, Hoffman-Censits J, Perez-Gracia JL, Dawson NA, van der Heijden MS, Dreicer R, Srinivas S, Retz MM, Joseph RW, Drakaki A, Vaishampayan UN, Sridhar SS, Quinn DI, Duran I, Shaffer DR, Eigl BJ, Grivas PD, Yu EY, Li S, Kadel EE 3rd, Boyd Z, Bourgon R, Hegde PS, Mariathasan S, Thastrom A, Abidoye OO, Fine GD, Bajorin DF; IMvigor210 Study Group. Atezolizumab as first-line treatment in cisplatin-ineligible patients with locally advanced and metastatic urothelial carcinoma: a single-arm, multicentre, phase 2 trial. Lancet. 2017 Jan 7;389(10064):67-76. doi: 10.1016/S0140-6736(16)32455-2. Epub 2016 Dec 8. PMID 27939400
- [Derived] Kim YS, Lee SI, Park SH, Park S, Hwang IG, Lee SC, Sun JM, Lee J, Lim HY. A Phase II Study of Weekly Docetaxel as Second-Line Chemotherapy in Patients With Metastatic Urothelial Carcinoma. Clin Genitourin Cancer. 2016 Feb;14(1):76-81. doi: 10.1016/j.clgc.2015.09.008. Epub 2015 Sep 25. PMID 26454620

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel): Participants randomized to the chemotherapy arm received vinflunine, paclitaxel, or docetaxel per the investigators choice. Vinflunine 320 milligrams per square meter (mg/m^2), paclitaxel 175 mg/m^2, or docetaxel 75 mg/m^2 were administered intravenously on Day 1 of each 21-day cycle until disease progression per standard RECIST v1.1 or unacceptable toxicity.
- Atezolizumab: Atezolizumab was administered intravenously at a fixed dose of 1200 milligrams (mg) on Day 1 of each 21-day cycle. Participants received atezolizumab as long as they continued to experience clinical benefit in the opinion of the investigator until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator.
Period: Overall Study
Arm/Group | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab
Started | 464 | 467
Received Treatment | 443 | 459
Completed | 0 (Participants still on chemotherapy were discontinued where that treatment was available locally.) | 0 (Participants still receiving atezolizumab had opportunity to continue treatment in extension study.)
Not Completed | 464 | 467
Not completed — Withdrawal by Subject | 28 | 11
Not completed — Lost to Follow-up | 4 | 6
Not completed — Death | 397 | 385
Not completed — Study Terminated By Sponsor | 35 | 64
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab | Total
Number analyzed (Participants) | 464 | 467 | 931
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (9.3) | 65.9 (9.6) | 66.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 110 | 213
  Male | 361 | 357 | 718
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 13 | 29
  Not Hispanic or Latino | 368 | 363 | 731
  Unknown or Not Reported | 80 | 91 | 171
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 55 | 63 | 118
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 336 | 335 | 671
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 70 | 68 | 138

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as time from randomization to death from any cause.
Time Frame: Between randomization and death due to any cause, up to approximately 25 months after first participant enrolled
Population: Intent To Treat (ITT) was defined as all randomized participants, irrespective of whether the assigned treatment was actually received.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- IC2/3 Chemotherapy; IC2/3 Atezolizumab: PD-L1 immunohistochemistry (IHC) score of IC2/3
- IC1/2/3 Chemotherapy; IC1/2/3 Atezolizumab: PD-L1 immunohistochemistry (IHC) score of IC1/2/3
Arm/Group | IC2/3 Chemotherapy | IC2/3 Atezolizumab | IC1/2/3 Chemotherapy | IC1/2/3 Atezolizumab | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab
Number analyzed (Participants) | 118 | 116 | 309 | 316 | 464 | 467
Months | 10.6 [8.4 to 12.2] | 11.1 [8.6 to 15.5] | 8.2 [7.4 to 9.5] | 8.9 [8.2 to 10.9] | 8.0 [7.2 to 8.6] | 8.6 [7.8 to 9.6]
Statistical Analysis 1: Comparison: IC2/3 Chemotherapy vs IC2/3 Atezolizumab; Test type: Superiority; p = 0.4134, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.63 to 1.21]
Statistical Analysis 2: Comparison: IC1/2/3 Chemotherapy vs IC1/2/3 Atezolizumab; Test type: Superiority; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.71 to 1.05]
Statistical Analysis 3: Comparison: Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) vs Atezolizumab; Test type: Superiority; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.73 to 0.99]

2. Secondary Outcome: Progression-free Survival (PFS) as Determined by the Investigator With Use of RECIST v1.1
Description: PFS was defined as the time between the date of randomization and the date of first documented progression of disease (PD) or death, whichever occurred first. PD was determined on the basis of investigator assessment with use of RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters had to demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: Up to approximately 25 months after first participant enrolled
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab | IC2/3 Chemotherapy | IC2/3 Atezolizumab | IC1/2/3 Chemotherapy | IC1/2/3 Atezolizumab
Number analyzed (Participants) | 464 | 467 | 118 | 116 | 309 | 316
months | 4.0 [3.4 to 4.2] | 2.1 [2.1 to 2.2] | 4.2 [3.7 to 5.0] | 2.4 [2.1 to 4.2] | 4.1 [3.6 to 4.2] | 2.1 [2.1 to 2.2]

3. Secondary Outcome: Unconfirmed Duration of Response (DOR) as Determined by the Investigator With Use of RECIST v1.1
Description: DOR was defined as the time from first occurrence of a CR or PR, whichever came first, to first documented PD or death, whichever occurred first. Disease progression was determined on the basis of investigator assessment with use of RECIST v1.1. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 mm.
Time Frame: Up to approximately 25 months after first participant enrolled
Population: DOR analyses was performed on the subset of patients who achieved an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab | IC2/3 Chemotherapy | IC2/3 Atezolizumab | IC1/2/3 Chemotherapy | IC1/2/3 Atezolizumab
Number analyzed (Participants) | 96 | 71 | 34 | 30 | 68 | 51
months | 5.3 [4.2 to 6.3] | 21.7 [9.9 to 21.7] | 6.4 [4.2 to 8.3] | 13.0 [6.6 to NA] — The DOR data was not mature at the time of clinical cutoff (i.e., majority of the responders are still ongoing), so the upper confidence interval was not estimable. | 5.5 [4.2 to 7.4] | 13 [6.9 to NA] — The DOR data was not mature at the time of clinical cutoff (i.e., majority of the responders are still ongoing), so the upper confidence interval was not estimable.

4. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to approximately 46 months after first participant enrolled
Population: Safety analyses was performed on all randomized patients who received any amount of study treatment, with patients grouped according to whether any amount of atezolizumab was received including the case when atezolizumab was received in error.
Measure: Number; unit: percentage
Arm/Group | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab | IC2/3 Chemotherapy | IC2/3 Atezolizumab | IC1/2/3 Chemotherapy | IC1/2/3 Atezolizumab
Number analyzed (Participants) | 443 | 459 | 112 | 114 | 297 | 312
percentage | 98.2 | 95.0 | 98.2 | 96.5 | 98.7 | 96.2

5. Secondary Outcome: Percentage of Participants With Post-Baseline Anti-therapeutic Antibodies (ATA) to Atezolizumab
Description: Participants were considered post-baseline ATA positive if they had post-baseline ATAs to Atezolizumab that were treatment-induced or treatment-enhanced. Participants had treatment-induced ATAs if they had a baseline-negative ATA result and developed ATAs at any time after initial drug administration. Participants had treatment-enhanced ATAs if they had a baseline-positive ATA result that showed an enhanced signal that was >/= 0.60 titer units at any time after initial drug initiation.
Time Frame: Predose (0 hours) on Day 1 of Cycles 1, 2, 3, 4 and every 8 cycles thereafter; at treatment discontinuation (up to 25 months); at 120 days after last dose of atezolizumab (up to 25 months; each cycle is 21 days)
Population: ATA evaluable population is defined as patients who received atezolizumab treatment and had at least one post-treatment ATA result.
Measure: Number; unit: percentage of participants
Groups:
- IC1/2/3 Atezolizumab; IC2/3 Atezolizumab: PD-L1 immunohistochemistry (IHC) score of IC2/3
Arm/Group | Atezolizumab | IC1/2/3 Atezolizumab | IC2/3 Atezolizumab
Number analyzed (Participants) | 427 | 289 | 106
percentage of participants | 33.3 | 35.0 | 33.0

6. Secondary Outcome: Minimum Observed Serum Atezolizumab Concentration (Cmin)
Description: Cmin was measured for all participants that received at least one dose of Atezolizumab.
Time Frame: as for outcome 5
Population: The PK-evaluable population is defined as patients who received atezolizumab treatment and had at least one measureable PK concentration.
Measure: Geometric Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab
Number analyzed (Participants) | 467
mcg/mL
  Cycle 2, day 1: number analyzed (Participants) | 399
  Cycle 2, day 1 | 67.5 (29.1)
  Cycle 3, day 1: number analyzed (Participants) | 341
  Cycle 3, day 1 | 95.1 (46.5)
  Cycle 4, day 1: number analyzed (Participants) | 259
  Cycle 4, day 1 | 122 (56.9)
  Cycle 8, day 1: number analyzed (Participants) | 156
  Cycle 8, day 1 | 159 (72.4)
  Cycle 16, day 1: number analyzed (Participants) | 79
  Cycle 16, day 1 | 190 (94.7)
  Cycle 24, day 1: number analyzed (Participants) | 30
  Cycle 24, day 1 | 190 (98.7)
  Cycle 32, day 1: number analyzed (Participants) | 8
  Cycle 32, day 1 | 223 (87.4)

7. Secondary Outcome: Percentage of Participants With Unconfirmed Objective Response Rate (ORR) as Determined by the Investigator With Use of Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1)
Description: ORR was defined as the percentage of participants, who had an objective response. Objective response was defined as either a complete response (CR) or partial response (PR) as determined by the investigator with use of Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1). Objective response in this study did not need to be a confirmed response. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. ORR=CR+PR
Time Frame: Up to approximately 25 months after first participant enrolled
Population: ORR analyses was performed on all randomized patients who had measureable disease at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab | IC2/3 Chemotherapy | IC2/3 Atezolizumab | IC1/2/3 Chemotherapy | IC1/2/3 Atezolizumab
Number analyzed (Participants) | 461 | 462 | 116 | 113 | 306 | 312
Percentage of participants | 20.8 [17.21 to 24.82] | 15.4 [12.20 to 18.99] | 29.3 [21.23 to 38.48] | 26.5 [18.68 to 35.68] | 22.2 [17.69 to 27.30] | 16.3 [12.42 to 20.93]

8. Secondary Outcome: Maximum Observed Serum Atezolizumab Concentration (Cmax)
Description: Cmax was measured for all participants that received at least one dose of Atezolizumab.
Time Frame: 30 minutes post dose on Day 1 of Cycles 1
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab
Number analyzed (Participants) | 467
mcg/mL | 334 (125)

9. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire Core 30 (QLQ-C30) Score: Global Health Status Scale
Description: The EORTC QLQ-C30 includes five functional scales (physical, role, cognitive, emotional, social); a global health status (GHS)/quality of life (QoL) scale; and items measuring fatigue, pain, nausea and vomiting, dyspnea, appetite loss, sleep disturbance, constipation, diarrhea, and financial difficulties. The score range for each scale and single-item measure is 0 to 100, where higher scores indicate a higher response level (i.e., better functioning, better QoL, worse symptoms). Key scales included physical functioning, and fatigue, and GHS.
Time Frame: Cycle 1 Day 1 (prior to any health care interaction), on Day 1 of each subsequent cycle, and at 30 days after the last treatment dose (Up to approximately 25 months; each cycle is 21 days)
Population: All randomized patients with non-missing baseline assessment and at least one non-missing post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units of a scale
Arm/Group | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab
Number analyzed (Participants) | 381 | 408
units of a scale
  Baseline (Cycle 1, Day 1): number analyzed (Participants) | 380 | 407
  Baseline (Cycle 1, Day 1) | 61.49 (22.30) | 64.19 (21.72)
  Change from baseline: Cycle 2, Day 1: number analyzed (Participants) | 349 | 379
  Change from baseline: Cycle 2, Day 1 | -5.47 (20.02) | -6.18 (20.07)
  Change from baseline: Cycle 3, Day 1: number analyzed (Participants) | 299 | 328
  Change from baseline: Cycle 3, Day 1 | -3.76 (22.34) | -4.67 (20.89)
  Change from baseline: Cycle 4, Day 1: number analyzed (Participants) | 203 | 250
  Change from baseline: Cycle 4, Day 1 | -1.48 (19.71) | -0.53 (20.23)
  Change from baseline: Cycle 12, Day 1: number analyzed (Participants) | 38 | 104
  Change from baseline: Cycle 12, Day 1 | -3.95 (24.33) | -0.56 (22.31)
  Change from baseline: Cycle 20, Day 1: number analyzed (Participants) | 11 | 68
  Change from baseline: Cycle 20, Day 1 | -2.27 (16.28) | 1.10 (21.88)
  Change from baseline: Cycle 28, Day 1: number analyzed (Participants) | 5 | 19
  Change from baseline: Cycle 28, Day 1 | -11.67 (7.45) | -5.26 (33.82)
  Change from baseline:Treatment Discont. Visit: number analyzed (Participants) | 267 | 200
  Change from baseline:Treatment Discont. Visit | -10.77 (24.15) | -16.71 (24.39)

10. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire Core 30 (QLQ-C30) Score: Physical Functioning Scale
Description: as for outcome 9
Time Frame: as for outcome 9
Population: All randomized patients with non-missing baseline assessment and at least one non-missing post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units of a scale
Arm/Group | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab
Number analyzed (Participants) | 381 | 408
units of a scale
  Baseline (Cycle 1, Day 1) | 74.23 (22.55) | 76.37 (19.66)
  Change from baseline: Cycle 2, Day 1: number analyzed (Participants) | 351 | 385
  Change from baseline: Cycle 2, Day 1 | -4.80 (15.70) | -7.56 (18.24)
  Change from baseline: Cycle 3, Day 1: number analyzed (Participants) | 303 | 331
  Change from baseline: Cycle 3, Day 1 | -5.64 (17.37) | -7.06 (19.62)
  Change from baseline: Cycle 4, Day 1: number analyzed (Participants) | 202 | 254
  Change from baseline: Cycle 4, Day 1 | -4.41 (16.25) | -3.81 (17.49)
  Change from baseline: Cycle 12, Day 1: number analyzed (Participants) | 39 | 105
  Change from baseline: Cycle 12, Day 1 | -6.97 (20.20) | 0.89 (16.23)
  Change from baseline: Cycle 20, Day 1: number analyzed (Participants) | 11 | 69
  Change from baseline: Cycle 20, Day 1 | -3.03 (11.30) | 3.48 (13.56)
  Change from baseline: Cycle 28, Day 1: number analyzed (Participants) | 5 | 19
  Change from baseline: Cycle 28, Day 1 | -18.67 (24.68) | 3.51 (20.53)
  Change from baseline: Treatment Discont. Visit: number analyzed (Participants) | 267 | 201
  Change from baseline: Treatment Discont. Visit | -15.58 (25.67) | -20.19 (25.52)

11. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire Core 30 (QLQ-C30) Score: Fatigue Symptom Scale
Description: as for outcome 9
Time Frame: as for outcome 9
Population: All randomized patients with non-missing baseline assessment and at least one non-missing post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units of a scale
Arm/Group | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab
Number analyzed (Participants) | 381 | 408
units of a scale
  Fatigue Symptom: Baseline (Cycle 1, Day 1) | 34.67 (26.66) | 32.87 (23.88)
  Fatigue Symptom: Cycle 2, Day 1: number analyzed (Participants) | 350 | 385
  Fatigue Symptom: Cycle 2, Day 1 | 10.71 (23.13) | 10.56 (21.82)
  Change from baseline: Cycle 3, Day 1: number analyzed (Participants) | 302 | 329
  Change from baseline: Cycle 3, Day 1 | 11.04 (25.48) | 9.41 (24.80)
  Change from baseline: Cycle 4, Day 1: number analyzed (Participants) | 202 | 254
  Change from baseline: Cycle 4, Day 1 | 7.48 (22.63) | 3.67 (23.57)
  Change from baseline: Cycle 12, Day 1: number analyzed (Participants) | 39 | 105
  Change from baseline: Cycle 12, Day 1 | 5.70 (27.44) | -0.95 (23.27)
  Change from baseline: Cycle 20, Day 1: number analyzed (Participants) | 11 | 69
  Change from baseline: Cycle 20, Day 1 | 11.11 (28.97) | -8.05 (21.97)
  Change from baseline: Cycle 28, Day 1: number analyzed (Participants) | 5 | 19
  Change from baseline: Cycle 28, Day 1 | 15.56 (16.85) | -12.28 (28.42)
  Change from baseline: Treatment Discont. Visit: number analyzed (Participants) | 267 | 201
  Change from baseline: Treatment Discont. Visit | 17.27 (28.15) | 19.60 (25.95)

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 8 Nov 2018 (up to 46 months)
Groups:
- Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel): Participants randomized to the chemotherapy arm will receive vinflunine, paclitaxel, or docetaxel per the investigator's choice. Vinflunine 320 milligrams per square meter (mg/m^2), paclitaxel 175 mg/m^2, or docetaxel 75 mg/m^2 will be administered intravenously on Day 1 of each 21-day cycle until disease progression per standard RECIST v1.1 or unacceptable toxicity.
Arm/Group | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 393/443 | 379/459
Serious Adverse Events (participants affected / at risk) | 189/443 | 192/459
Other Adverse Events (participants affected / at risk) | 417/443 | 413/459
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) (N=443) | Atezolizumab (N=459)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 9 (9)
Bone Marrow Failure (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 22 (25) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 14 (15) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Acute Coronary Syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 1 (2)
Macular Fibrosis (Eye disorders) | 0 (0) | 1 (1)
Papilloedema (Eye disorders) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 9 (9) | 5 (5)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 3 (3)
Anal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Autoimmune Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 20 (23) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 6 (6)
Duodenal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 6 (6) | 1 (2)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 (4) | 1 (1)
Subileus (Gastrointestinal disorders) | 4 (4) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5)
Death (General disorders) | 2 (2) | 3 (3)
Fatigue (General disorders) | 5 (6) | 4 (4)
General Physical Health Deterioration (General disorders) | 4 (4) | 2 (2)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1)
Injection Site Reaction (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 2 (2) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Obstruction (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (4) | 3 (3)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 17 (18)
Strangulated Hernia (General disorders) | 1 (1) | 1 (1)
Autoimmune Hepatitis (Hepatobiliary disorders) | 0 (0) | 4 (5)
Biliary Dilation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatocellular Injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Arthritis Infective (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 2 (2)
Enterococcal Infection (Infections and infestations) | 1 (2) | 0 (0)
Enterococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 1 (3)
Escherichia Infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella Infection (Infections and infestations) | 0 (0) | 2 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2)
Meningoencephalitis Viral (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic Infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Ophthalmic Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 4 (5)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 15 (16) | 8 (8)
Septic Shock (Infections and infestations) | 2 (2) | 2 (2)
Spinal Cord Infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 1 (1)
Toxic Shock Syndrome (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 14 (17) | 21 (25)
Urinary Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 12 (12) | 2 (2)
Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma Site Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Urostomy Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1) | 2 (2)
Blood Creatinine Increased (Investigations) | 1 (1) | 1 (1)
Liver Function Test Abnormal (Investigations) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 4 (4) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mantle Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumor Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain Oedema (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 2 (2)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Device Dislocation (Product Issues) | 1 (1) | 0 (0)
Device Occlusion (Product Issues) | 3 (5) | 1 (2)
Completed Suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 6 (6) | 11 (12)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder Perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Tamponade (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 7 (9) | 10 (19)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 3 (3)
Postrenal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 5 (5) | 4 (4)
Renal Haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral Haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 6 (6)
Urinary Tract Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 4 (4)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Thrombophlebitis (Vascular disorders) | 3 (3) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2)
Unevaluable Event (General disorders) | 0 (0) | 1 (1)
Escherichia Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pyonephrosis (Infections and infestations) | 0 (0) | 1 (1)
Vascular Device Infection (Infections and infestations) | 4 (4) | 0 (0)
Skin Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 1 (1)
Genital Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Internal Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (Vinflunine, Paclitaxel, or Docetaxel) (N=443) | Atezolizumab (N=459)
Anaemia (Blood and lymphatic system disorders) | 124 (142) | 90 (94)
Neutropenia (Blood and lymphatic system disorders) | 57 (75) | 5 (6)
Abdominal Pain (Gastrointestinal disorders) | 58 (63) | 52 (60)
Abdominal Pain Upper (Gastrointestinal disorders) | 27 (32) | 23 (23)
Constipation (Gastrointestinal disorders) | 163 (221) | 131 (147)
Diarrhoea (Gastrointestinal disorders) | 94 (115) | 97 (145)
Dry Mouth (Gastrointestinal disorders) | 8 (8) | 30 (36)
Nausea (Gastrointestinal disorders) | 137 (171) | 106 (124)
Stomatitis (Gastrointestinal disorders) | 35 (41) | 13 (16)
Vomiting (Gastrointestinal disorders) | 81 (108) | 55 (67)
Asthenia (General disorders) | 107 (144) | 92 (108)
Fatigue (General disorders) | 136 (162) | 129 (153)
Mucosal Inflammation (General disorders) | 47 (64) | 27 (30)
Oedema Peripheral (General disorders) | 36 (43) | 52 (59)
Pain (General disorders) | 31 (34) | 24 (24)
Pyrexia (General disorders) | 62 (76) | 93 (128)
Nasopharyngitis (Infections and infestations) | 11 (15) | 27 (43)
Urinary Tract Infection (Infections and infestations) | 58 (76) | 84 (141)
Blood Creatinine Increased (Investigations) | 11 (12) | 36 (38)
Neutrophil Count Decreased (Investigations) | 26 (49) | 0 (0)
Weight Decreased (Investigations) | 45 (46) | 47 (47)
Decreased Appetite (Metabolism and nutrition disorders) | 113 (136) | 135 (147)
Hypokalaemia (Metabolism and nutrition disorders) | 23 (26) | 16 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 60 (79) | 47 (66)
Back Pain (Musculoskeletal and connective tissue disorders) | 51 (53) | 80 (95)
Bone Pain (Musculoskeletal and connective tissue disorders) | 24 (28) | 24 (27)
Myalgia (Musculoskeletal and connective tissue disorders) | 55 (68) | 25 (27)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 48 (55) | 37 (46)
Dizziness (Nervous system disorders) | 30 (32) | 29 (29)
Dysgeusia (Nervous system disorders) | 25 (27) | 12 (14)
Headache (Nervous system disorders) | 26 (35) | 38 (44)
Neuropathy Peripheral (Nervous system disorders) | 55 (67) | 8 (9)
Paraesthesia (Nervous system disorders) | 29 (32) | 18 (18)
Peripheral Sensory Neuropathy (Nervous system disorders) | 41 (43) | 6 (7)
Anxiety (Psychiatric disorders) | 24 (24) | 27 (27)
Insomnia (Psychiatric disorders) | 42 (42) | 45 (48)
Haematuria (Renal and urinary disorders) | 26 (32) | 45 (60)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (36) | 59 (69)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 (50) | 62 (70)
Alopecia (Skin and subcutaneous tissue disorders) | 125 (127) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (27) | 64 (86)
Rash (Skin and subcutaneous tissue disorders) | 28 (37) | 54 (72)
Hypertension (Vascular disorders) | 20 (22) | 23 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT02302807/Prot_SAP_001.pdf